CLINICAL TRIAL: NCT06167993
Title: Effect of Complex Decongestive Physiotherapy Applied After Lymphovenous Anastomosis Surgery on Extremity Volume, Quality of Life and Patient Satisfaction (Randomized Controlled Study)
Brief Title: Complex Decongestive Physiotherapy Applied After Lymphovenous Anastomosis Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, hanife dogan, Principal Investigator, Necmettin Erbakan University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: hdogan
Record Dates: First submitted 2023-11-20; First posted 2023-12-13 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Lymphedema; Cancer
MeSH Terms: conditions — Lymphedema; Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group receiving CDP in patients who underwent LVA (Experimental): LVA: Group that underwent lymphovenous anastomosis surgery and CDP applied groups CDP:Complex Decongestive Physiotherapy
  Interventions: Behavioral: Complex Decongestive Physiotherapy
- Group receiving CDP after lymphedema (Active Comparator): Only CDP applied groups
  Interventions: Behavioral: Complex Decongestive Physiotherapy

INTERVENTIONS:
Behavioral: Complex Decongestive Physiotherapy — Complex Decongestive Physiotherapy; It consists of manual therapy, skin care, compression therapy and therapeutic exercise.

SUMMARY:
Type of this study: Prospective randomized controlled study. The aim of our study is to compare patients with lymphedema who have undergone lymphovenous anastomosis surgery receiving Complex Decongestive Physiotherapy (CDP), patients with lymphedema who have not undergone surgery who receive Complex Decongestive Physiotherapy, in terms of Extremity Volume, Quality of Life and Patient Satisfaction.

26 volunteers will be included in the study as patients with lymphedema who have undergone lymphovenous anastomosis surgery and KBF (n=13), only KBF (n=13), application groups. How effective is lymphovenous anastomosis surgery and KBF or only CDP acutely in the treatment of lymhedema?

DETAILED DESCRIPTION:
Lymphedema (LE) is a chronic and progressive condition that occurs as a result of abnormal accumulation of protein-rich fluid in the interstitial space due to inadequate lymphatic drainage. The gold standard treatment program among physiotherapy applications is the Complex Decongestive Physiotherapy application. It consists of four basic components; Manual Lymph Drainage, Skin Care, Compression Therapy, Therapeutic Exercise. All patients will receive the treatment phase of KBF for 20 sessions, 5 days a week: Treatment; The 45-minute MLD consists of skin care, compression therapy with a short-draft bandage that they will then use for 23 hours a day, decongestive exercises and suggestions to facilitate venous and lymphatic flow. The effect of CDP will be compared in patients who have had lymphovenous anastomosis surgery and those who have not. Quality of life of patients related to lymphedema; Lymphedema Function, Disability and Health Questionnaire-Lower Extremity (LYMPH ICF-LL), satisfaction levels will be evaluated with the Visual analog scale, and the amount of edema will be evaluated with circumference measurement.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65,
* Having unilateral lower extremity or upper extremity lymphedema,
* Being diagnosed with Stage 2 and 3 lymphedema,
* Receiving lymphedema therapy for the first time,
* Adjuvant chemotherapy for gynecological cancer,
* Having completed radiation and surgical treatment at least 3 months and at most 5 years ago,
* Patients with lymph vessels seen on lymphangiography,
* Patients who have undergone LVA surgery and 1 month has passed since the surgery date
* No evidence of disease recurrence at last follow-up visit and
* Individuals willing to participate in the study

Exclusion Criteria:

* Those who do not volunteer to participate in the study,
* Those with bilateral lower extremity lymphedema,
* Having upper or lower extremity edema due to systemic disease,
* Those with active infection,
* Patients more than 1.5 months after LVA surgery
* Known to have mental and cognitive disorders
* Those who were unable to communicate and cooperate were not included.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Tape Measure | 5 months
  Extremity Volume; In calculating the circumference measurements of the lower and upper extremities, the circumference of the healthy and diseased extremities is measured at 4 cm intervals with the help of a tape measure. These circumference measurements (thickest and thinnest circumference measurement values) are then converted to volumetric measurements using the Frustum Formula.

SECONDARY OUTCOMES:
Lymphedema Function, Disability and Health Questionnaire-Lower Extremity (LYMPH ICF-LL) Scale | 5 months
  Evaluates patients' quality of life related to lymphedema.
Visual Analogue Scale (VAS) | 5 months
  VAS: A 10 cm visual analogue scale was used to evaluate the patients' satisfaction levels with the physiotherapy they received. The same evaluation was repeated before and after treatment. The patient will be asked to mark a field between the highest value of satisfaction level, 10, and the lowest value, "0".

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Bilsev İnce, Konya
  - Hanife Dogan, Konya

IPD SHARING:
Plan to Share IPD: No